CLINICAL TRIAL: NCT03010137
Title: Incisional Negative Pressure Wound Therapy in High Risk Patients Undergoing Panniculectomy: A Prospective Randomized Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of staff resources to properly consent and enroll patients into the study.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 801708
Record Dates: First submitted 2017-01-03; First posted 2017-01-04 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Complications Wounds; Negative Pressure Wound Therapy; Wound Healing Delayed; Incisional; Panniculectomy; Incisional Negative Pressure Wound Therapy; Incisional Vac; Wound Vac; Obese; Renal Failure; Kidney Transplant; Complications; Wound Healing Complication
MeSH Terms: conditions — Surgical Wound; Obesity; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Closure (Placebo Comparator): After surgical closure is complete, the patient receives standard of care operative incision treatment (dermabond/topical skin adhesive).
  Interventions: Procedure: Standard Closure with Skin Glue; Device: Dermabond
- Incisional Negative Pressure Wound Therapy (Active Comparator): After surgical closure is complete, an incisional negative pressure wound therapy device is applied to the incision in its entirety. This device is placed on the wound, sterilely, in the operating room, at the conclusion of the procedure. The incisional negative pressure wound therapy device is to remain in place for 7 days, and is removed in clinic after completion.
  Interventions: Procedure: Incisional Negative Pressure Wound Therapy; Device: PICO (Smith&Nephew)

INTERVENTIONS:
Procedure: Incisional Negative Pressure Wound Therapy
  Arms: Incisional Negative Pressure Wound Therapy
Procedure: Standard Closure with Skin Glue
  Arms: Standard Closure
Device: PICO (Smith&Nephew) — Off the shelf, disposable negative pressure wound therapy device. Contains sterile dressing as well as an attached small (pager sized) suction device/canister.
  Arms: Incisional Negative Pressure Wound Therapy
Device: Dermabond — Final wound closure with skin glue.
  Arms: Standard Closure

SUMMARY:
Incisional negative pressure therapy (INPWT) has previously been shown in certain patient populations to decrease wound healing complications, decrease the rate of hematomas and seromas, as well as have better scar quality. We have found a group of patients, those who have panniculectomies in preparation for renal transplant, with significantly higher rates of wound healing complications. We believe the best way to demonstrate benefits of incisional negative pressure wound therapy will be in this group of patients known to have significantly higher rates of wound complications.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing panniculectomy in preparation for renal transplantation at the University of California Davis Medical Center. Patients who are entered into the trial and have 30 days of follow up, and those in the INPWT study arm who successfully complete 7 days of treatment, will be included.

Exclusion Criteria:

* All patients who previously demonstrated a hypersensitivity reaction to adhesives and qualify for panniculectomy in preparation for renal transplantation, or all patients who are undergoing panniculectomy for reasons other than in preparation for renal transplantation (i.e. after massive weight loss or for cosmetic reasons). Patients who do not complete the duration of treatment of negative pressure wound therapy (7 days), or patients who do not follow up for a minimum of 30 days from the date of surgery will be excluded. Adults unable to consent, infants, children, teenagers, pregnant patients and prisoners will be excluded. It is also extremely unlikely, based on our study population, that we will encounter any of these patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12; Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Wong, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Closure: After surgical closure is complete, the patient receives standard of care operative incision treatment (dermabond/topical skin adhesive).
  Standard Closure with Skin Glue
  Dermabond: Final wound closure with skin glue.
- Incisional Negative Pressure Wound Therapy: After surgical closure is complete, an incisional negative pressure wound therapy device is applied to the incision in its entirety. This device is placed on the wound, sterilely, in the operating room, at the conclusion of the procedure. The incisional negative pressure wound therapy device is to remain in place for 7 days, and is removed in clinic after completion.
  Incisional Negative Pressure Wound Therapy
  PICO (Smith&Nephew): Off the shelf, disposable negative pressure wound therapy device. Contains sterile dressing as well as an attached small (pager sized) suction device/canister.
Period: Overall Study
Arm/Group | Standard Closure | Incisional Negative Pressure Wound Therapy
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Closure | Incisional Negative Pressure Wound Therapy | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 13 | 28
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (8.6) | 57 (10) | 55.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Major Wound Healing Complications
Description: Abscess, Hematoma or any wound complication requiring return to the operating room.
Time Frame: Up to 3 months after operation
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Closure | Incisional Negative Pressure Wound Therapy
Number analyzed (Participants) | 15 | 15
Participants | 5 | 3

2. Primary Outcome: Minor Wound Healing Complications
Description: Cellulitis, Seroma, Superficial Wound Separation
Time Frame: Up to 3 months after operation
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Closure | Incisional Negative Pressure Wound Therapy
Number analyzed (Participants) | 15 | 15
Participants | 3 | 2

3. Secondary Outcome: Time to Drain Removal
Description: Time to final drain removal after the operation
Time Frame: Up to 3 months after operation
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard Closure | Incisional Negative Pressure Wound Therapy
Number analyzed (Participants) | 15 | 15
days | 29 (14.1) | 24 (13.5)

4. Other Pre Specified Outcome: Scarring
Description: Will assess using Vancouver Scar Scale
Time Frame: data not collected due to early termination
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Pain Score Self Reported by the Patient After Surgery
Description: Assess via a visual analog scale at specified intervals
Time Frame: data not collected due to early termination
Population: Unable to perform final analysis due to early closure of the study
Arm/Group | Standard Closure | Incisional Negative Pressure Wound Therapy
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Quality of Life as Measured by SF-36 Validated Survey
Description: Assess via SF-36 validated survey at specified intervals
Time Frame: data not collected due to early termination
Population: unable to perform final analysis due to early termination of study
Arm/Group | Standard Closure | Incisional Negative Pressure Wound Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months period following panniculectomy surgery
Arm/Group | Standard Closure | Incisional Negative Pressure Wound Therapy
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-10-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT03010137/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT03010137/ICF_001.pdf